CLINICAL TRIAL: NCT01894620
Title: Investigating the Effect of Repetitive Transcranial Magnetic Stimulation as a Treatment for Alzheimer's Disease and on Sleep Quality
Brief Title: The Effect of rTMS Treatment on Alzheimer's and Sleep Quality
Acronym: rTMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Zahra Kazem-Moussavi (Other)
Responsible Party: Sponsor-Investigator, Dr. Zahra Kazem-Moussavi, Professor, University of Manitoba
Organization: University of Manitoba (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: B2012:76
Record Dates: First submitted 2013-07-03; First posted 2013-07-10 (Estimated); Results first posted 2018-02-12 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's; rTMS; sleep quality; dementia; memory
MeSH Terms: conditions — Alzheimer Disease; Sleep Initiation and Maintenance Disorders; Dementia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- rTMS with sham coil (Placebo Comparator): rTMS real-sham and rTMS sham-real interventions. Each patient will receive both real and sham treatment in two different blocks of time. The assessments after the sham treatment will serve as placebo effect compared to those after real treatment.
  Interventions: Device: rTMS real-sham; Device: rTMS sham-real
- rTMS with real coil (Active Comparator): rTMS real-sham and rTMS sham-real interventions. Each patient will receive both real and sham treatment in two different blocks of time. The assessments after the sham treatment will serve as placebo effect compared to those after real treatment.
  Interventions: Device: rTMS real-sham; Device: rTMS sham-real

INTERVENTIONS:
Device: rTMS real-sham — In this intervention patients receive 4 weeks of rTMS treatment with real coil and then 4 weeks of treatment with sham coil; there will be 4 weeks of break between the two blocks of treatment.
Device: rTMS sham-real — In this intervention patients receive 4 weeks of rTMS treatment with sham coil and then 4 weeks of treatment with real coil; there will be 4 weeks of break between the two blocks of treatment.

SUMMARY:
This research is being conducted to study whether rTMS (repetitive Transcranial Magnetic Stimulation) could be potentially used as a treatment for Alzheimer's disease. rTMS is a technique that stimulates the brain by rapidly switching a magnetic field in a coil placed over your head. Prior to rTMS, single pulse TMS will be used to localize the specific brain region that we are interested in.

DETAILED DESCRIPTION:
Upon meeting the inclusion criteria and providing informed consent, each participant will complete a series of cognitive assessments and rTMS treatments at the TMS Lab at Riverview Health Center. Each treatment session will involve implementing rTMS, while the patient is involved in a cognitive exercise such as naming object or action. The study sessions will be scheduled as follows: Block 1: 5 days/week for two weeks followed by 2 days a week for 1 week, followed by once a week for 1 week (total of 13 treatments); Pause: 4 weeks of no treatment; and Block 2: another 13 sessions of treatment with the same pattern as Block 1. One of these two sets of treatment (Block 1 or Block 2) will be sham and one will be real. Sham treatment sessions are identical to real treatment sessions, except that there is no magnetic stimulation. Patients will be randomly assigned to receive either sham or real treatment first. The purpose of sham treatment is to have a control group data that the plausible improvement as a result of rTMS can be compared to. By designing two sets of sham-real or real-sham treatment sessions, every participant will receive a real treatment, while we will also have control data.

The cognitive assessments will be done at the baseline, and then on weekly basis. A subgroup of the study population will be recruited for investigating the second objective: effect of rTMS on sleep quality. Those patients will be required to sign a second consent; then, the patients will go through full-night sleep study at Misericordia Health Center at the same time intervals as their cognitive assessments.

ELIGIBILITY:
Inclusion Criteria:

* Individuals must have a MoCA score between 5 and 26, indicating mild cognitive impairment or dementia.
* Participants must have probable early or moderate Alzheimer's disease as confirmed by their treating neurologist or psychiatrist, and/or by the co-investigators.

Exclusion Criteria:

* A recent (the last 3 months) history of stroke, recent (the last 3 months) head injury and loss of consciousness, any history of epilepsy, seizures, multiple sclerosis (MS), Amyotrophic Lateral Sclerosis (ALS), or Autism.
* Recent changes in medication (i.e. patients should be in a relatively stable phase of disease).
* The presence of metallic objects in the body; dental implants are fine but people with pacemakers are to be excluded; basically anything that is unsafe under MRI would be considered unsafe for TMS application.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2013-05; Primary Completion 2014-05 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zahra Kazem-Moussavi, Ph.D., Principal Investigator — University of Manitoba
Locations (2):
- Canada (2):
  - Misericordia Health Center, Winnipeg, Manitoba
  - Riverview Health Center, Winnipeg, Manitoba

RESULTS

PARTICIPANT FLOW:
Groups:
- rTMS Real-sham; rTMS Sham-real: rTMS real-sham and rTMS sham-real interventions. Each patient will receive both real and sham treatment in two different blocks of time. The assessments after the sham treatment will serve as placebo effect compared to those after real treatment.
  rTMS real-sham: In this intervention patients receive 4 weeks of rTMS treatment with real coil and then 4 weeks of treatment with sham coil; there will be 4 weeks of break between the two blocks of treatment.
  rTMS sham-real: In this intervention patients receive 4 weeks of rTMS treatment with sham coil and then 4 weeks of treatment with real coil; there will be 4 weeks of break between the two blocks of treatment.
Period: Overall Study
Arm/Group | rTMS Real-sham | rTMS Sham-real
Started | 6 | 5
Completed | 6 | 4
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | rTMS Real-sham | rTMS Sham-real | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 4 | 3 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.83 (10.48) | 68.25 (9.88) | 68.60 (9.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  Canada | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Cognitive Improvement Measured Using Montreal Cognitive Assessment (MoCA)
Description: We anticipate to see a cognitive improvement as measured by the Montreal Cognitive Assessment (MoCA) after two weeks of applying rTMS. This assessment tool gives a score from 0 to 30 points, with higher scores representing better cognitive ability.
Time Frame: Change between baseline and 2 weeks after the start of treatment
Population: Results are divided into the two treatment type groups (real vs. sham).
Measure: Mean (Standard Error); unit: MOCA score change at 2 weeks
Arm/Group | rTMS With Sham Coil | rTMS With Real Coil
Number analyzed (Participants) | 10 | 10
MOCA score change at 2 weeks | -0.667 (1.116) | 1.8 (0.633)

2. Secondary Outcome: Improvement in Sleep Quality
Description: We anticipate to see an improvement on the sleep quality of the patients (assessed by EEG waves during sleep) after 4 weeks of rTMS treatment.
Time Frame: After four weeks after the start of treatment
Population: Note that this aspect of the study was not performed. Therefore, no data is available.
Arm/Group | rTMS Real-sham | rTMS Sham-real
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Full study (18 months)
Arm/Group | rTMS With Sham Coil | rTMS With Real Coil
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No